CLINICAL TRIAL: NCT03326167
Title: Determination of Coronary Flow Reserve by Dynamic Myocardial Perfusion Scintigraphy
Acronym: ERCAD
Status: Terminated | Type: Observational
Why Stopped: recruitment difficulty
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0259
Record Dates: First submitted 2017-10-26; First posted 2017-10-31 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with or suspected coronary heart disease
  Interventions: Other: Myocardial Perfusion Imaging by Single Photon Emission Computed Tomography (MPI SPECT)

INTERVENTIONS:
Other: Myocardial Perfusion Imaging by Single Photon Emission Computed Tomography (MPI SPECT) — Evaluation of the improvement of the sensitivity, in tri-truncular patients, provided by the estimation of the coronal reserve by territory, during the realization of a myocardial perfusion tomoscintigraphy on CZT camera dedicated to cardiology (Discovery NM 530 ).

SUMMARY:
Because of its availability, non-invasiveness, and high diagnostic performance, myocardial perfusion tomoscintigraphy has become a standard tool for the detection, characterization and monitoring of coronary artery disease. Standard analysis, based on the reversibility of regional myocardial hypoperfusion between stress (physiological or pharmacological) and rest, has good sensitivity and negative predictive value in the search for myocardial ischemia. However, two major obstacles persist. First, because of the relative nature of the normalization of cardiac activity, this approach may underestimate the extent of the damage, especially when the territory with the most activity is itself pathological. Thus myocardial perfusion scintigraphy can only detect 40 to 50% of tri-truncal patients. To overcome these disadvantages, several indexes have been proposed to improve the diagnostic performance of perfusion scintigraphy in multi-truncal patients based in particular on kinetic analysis. Secondly, the review does not provide any guarantee as to the quality and reproducibility of use of the coronal reserve during stress, in particular during submaximal stress tests and pharmacological stress, the latter being easily antagonized by xanthine derivatives contained in tea and coffee in particular (abstinence of at least 12 to 24 hours being recommended). In recent years and thanks to the advent of CZT semiconductor cameras dedicated to cardiology - to perform a dynamic tomographic acquisition - a study of the coronal reserve is feasible by perfusion tomoscintigraphy in current practice. This study of the coronary reserve mainly consists of a computer post-processing of the myocardial perfusion scintigraphy data and does not therefore require any additional irradiation (the only difference with respect to the old protocols is the start of the images at the time of publication. injection of the radiotracer). However, the diagnostic benefit gained from the coronary reserve study compared to conventional stress / rest perfusion scintigraphy has not been clearly studied, particularly in the multi-truncal patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients sent to the Nuclear Medicine Department as part of a functional evaluation by dynamic acquisition tomoscintigraphy and who will benefit from coronary angiography in the Louis Pradel Hospital hemodynamics department, depending on the results and the clinical context , outside of an emergency context.
* Patients who received the information and did not object to participate in the study

Exclusion Criteria:

* Patient with a contraindication to pharmacological stress by dipyridamole or regadenoson (acute coronary syndrome, acute pulmonary embolism, hypertension) severe pulmonary artery disease, acute aortic dissection, symptomatic aortic stenosis, hemodynamic instability, acute myocarditis, pericarditis or endocarditis, severe chronic obstructive pulmonary disease, uncompacted type III atrioventricular block, systolic pressure <90 mmHg, Recent ischemic stroke, hypersensitivity or allergy to active ingredients or excipients)
* Patients under 18 years of age
* Patients with atrial fibrillation complete arrhythmia (ACFA)
* Patients with a history of coronary bypass grafting.
* Patients whose clinical condition requires rapid management not allowing to wait for the completion of the exams
* Pregnancy and breast feeding
* Deprivation of civil rights (guardianship, guardianship, safeguard of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is conducted in adults with suspected coronary artery disease or coronary heart disease and referred for functional evaluation by perfusion scintigraphy with dynamic acquisition before coronary angiography.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-03-13 (Actual)

PRIMARY OUTCOMES:
Presence of significant stenosis in each of the three coronary areas | two weeks after MPI SPECT
  The gold standard will be provided by coronarography with Fractional Flow Reserve measurement during the angiographic procedure if necessary. Coronary stenosis with Fractional Flow Reserve <0.8 will be retained as positive

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine Nucléaire - Hôpital Louis Pradel - Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No